CLINICAL TRIAL: NCT04132206
Title: ScleroBiotique: Longitudinal Characterization of Microbial Signature in Systemic Sclerosis Patients
Brief Title: Longitudinal Characterization of Microbial Signature in Systemic Sclerosis Patients
Acronym: ScleroBiotique
Status: Recruiting | Type: Observational
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 18-30
Record Dates: First submitted 2019-10-08; First posted 2019-10-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A biological collection called "MEDIBIOTE 2" will be set up in parallel for all the participants in this study, This will be managed by the CRB-HE biobank.
  It will consist on stool-derived samples (DNA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ScS patients: Patients will provide two stool samples: one collected the day of inclusion and a second, six months later
  Interventions: Other: stool sampling
- Healthy subjects: Healthy subjects will provide one stool sample at inclusion.
  Interventions: Other: stool sampling

INTERVENTIONS:
Other: stool sampling — Participants will provide two stool samples: one collected the day of inclusion and a second, six months later

SUMMARY:
Today, the study of gut microbiota has taken a prominent place in several fields of medical research. Numerous experimental data in humans and animals suggest that an imbalance in the composition of the microbiota could contribute to the pathophysiology of systemic autoimmune diseases such as Systemic Sclerosis (SCS). A future exploration of the microbiota, a source of diagnostic and/or prognostic biomarkers, may be very useful for tomorrow's medicine by proposing therapeutic interventions based on the correction of possible imbalances in the intestinal flora. Studies of the human gut microbiota in patients with ScS are limited to low-impact investigations, due to the lack of data on the clinical and biological characterization of the patients studied, and to the absence of longitudinal studies in the same patient. For this reason, we are interested in exploring the intestinal microbiota of ScS patients in a comprehensive and longitudinal way.

DETAILED DESCRIPTION:
This is an explorative, prospective, monocentric open-label study qualified as interventional researches at minimal risks and constraints (called in French RIPH, category 2).

This is a study of the gut microbiota and its characteristics in ScS patients, compared to control subjects (without ScS or other chronic diseases), matched on age and sex.

Participants provided two stool samples: one collected the day of inclusion and a second, six months later.

In parallel with the microbiota analysis, a clinical (digestive and extra digestive signs, severity) and biological characterization of the ScS will be carried out by the team of internists. This medical evaluation will be completed by an interview with a dietician to inform about the participant's eating habits, and any changes in the 7 days preceding the stool collection.

Microbial profiles will be obtained from the sequencing data using the specialized tools DADA2 and Kraken.

The search of characteristic signature of ScS will be performed by comparing ScS patients and healthy controls using a discriminant linear analysis (LDA) using the specialized tool LEfSe Main objective is to identify, through longitudinal follow-up, significant differences in the composition of the intestinal microbiota of ScS patients and healthy control subjects (matched on age and sex) in order to define a microbial signature specific to the ScS.

Secondary objectives are to study the stability over time of the identified microbial signatures, and to determine a correlation between the composition of the microbiota obtained in the ScS patient and the severity of his symptoms (diffuse skin disease, pulmonary interstitial disease, digestive disease...)

ELIGIBILITY:
Inclusion Criteria:

For ScS patients:

1. Patients with ScS according to ACR criteria.
2. Patients over 18 years old.
3. Patients who have signed the consent to participate in this study.

For control subjects:

1. Persons without diagnosis of ScS or any other chronic disease.
2. Persons over 18 years old.
3. Persons who have signed the consent to participate in this study

Exclusion Criteria:

* 1. Persons with severe anemia (Hb < 7 g/dL). 2. Persons who cannot read French. 3. For control subjects: Persons with a particular symptom (as an example of digestive disorders), or under long-term treatment related to another pathology.

  4. Persons treated with antibiotics, probiotics, prebiotics or any other treatment that may disrupt the gut microbiota within two months before stool sampling.

  5. Persons referred to the article L1121-5 to 1121-8 of the Public health code, namely :
* Pregnant, women in labour and breastfeeding mothers.
* Persons deprived of their liberty by a judicial or administrative decision.
* Persons undergoing psychiatric follow-up.
* Minors
* Persons of full-age who are subject to a legal protection measure or who are unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ScS according to ACR criteria,and healthy volunteers without diagnosis of ScS or any other chronic disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
Differences on gut microbiota composition (bacterial populations) of ScS overtime, at different taxonomic levels (from phyla to species if technique allows) versus healthy controls. | 7 months
  The patient participation at the study will last 7 months, but healthy volunteers will provide stool sample only once at study entry and won't be followed after that.

CONTACTS AND LOCATIONS:
Overall Officials: Chloé STAVRIS, MD, Principal Investigator — Hôpital Européen Marseille
Locations (1):
- Hôpital Européen Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided